CLINICAL TRIAL: NCT02240290
Title: A Single-Center, Open-Label Study of Excretion Balance, Pharmacokinetics, and Metabolism of 14C-Labeled Tozadenant After 240 mg Single Oral Dose Administration in Healthy Male Subjects
Brief Title: Study to Evaluate the Absorption, Distribution, Break Down and Elimination and the Safety of 14C-Labeled Tozadenant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biotie Therapies Inc. (Industry)
Collaborators: PRA Health Sciences (Industry); Tandem Labs (Unknown); Xceleron Inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PD0026; 2013-002640-85 (EudraCT Number); NL46031.056.13 (Other: CCMO Netherlands)
Record Dates: First submitted 2014-08-25; First posted 2014-09-15 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2014-09

CONDITIONS: N/A, as Healthy Volunteers
Keywords: C14; Dosimetry; Mass balance; ADME
MeSH Terms: interventions — tozadenant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tozadenant (Experimental): A single dose of 240 mg tozadenant (four 60 mg tablets) and a 74 kBq (2 μCi) 14C-labeled tozadenant capsule will be administered with 240 mL of water.
  Interventions: Drug: tozadenant tablet; Drug: C14-tozadenant capsule

INTERVENTIONS:
Drug: tozadenant tablet — Active substance: tozadenant Pharmaceutical form: Tablet Concentration: 240 mg Route of Administration: Oral administration
Drug: C14-tozadenant capsule — Active substance: C14-tozadenant Pharmaceutical form: Capsule Concentration: 74 kBq (2 μCi) Route of administration: Oral administration

SUMMARY:
The purpose of the study is to investigate how tozadenant is absorbed, distributed, broken down and eliminated from the body. The compound to be administered will be radiolabeled. This enables the investigator to trace the compound in blood, urine, feces, expired air and track what happens to it.

DETAILED DESCRIPTION:
PD0026 is a Phase 1, single-center, open-label, single-dose study to investigate the absorption, distribution, metabolism, and excretion (ADME) of 14C-labeled tozadenant. The primary objective is to determine the mass balance and the pharmacokinetics (PK) of total radioactivity in 6 healthy male subjects following a single oral dose of 14C-labeled tozadenant. Secondary objectives are to determine the PK of Tozadenant, to identify and quantify metabolites of tozadenant, and to gain further information on the tolerability and safety of tozadenant.

The variables related to the radiocarbon activity include the total radioactivity concentration in whole blood and plasma; the total radioactivity excretion in urine, feces, and expired air; and the corresponding PK parameters.

The concentrations and the corresponding PK parameters of tozadenant over time will be determined in plasma, urine, and feces.

In addition, the metabolites of tozadenant will be identified and quantified. The safety and tolerability variables include adverse events (AEs), vital signs, physical examination, standard 12 lead electrocardiogram (ECG) intervals, and clinical laboratory results.

The study will consist of a Screening Period of up to 20 days (Days -21 to -2) and a Study Period of 15 days. Therefore, the maximum duration of participation from Screening until discharge from the clinic for a subject is 35 days.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male between the ages of 18 and 55 years inclusive; subject may be of any racial group
* Subject is informed and given ample time and opportunity to think about his participation and has signed and dated the Independent Ethics Committee (IEC) approved written Informed Consent form
* Subject is considered reliable and capable of adhering to the protocol, according to the judgment of the Investigator, and is capable of communicating satisfactorily with the Investigator and complying with all study requirements
* Subject has a body mass index (BMI) between 18 to 30 kg/m², inclusive, and weighs at least 50 kg
* In the opinion of the Investigator, determined on the basis of the medical history and a general clinical examination at Screening, the subject has no clinically relevant cardiovascular, renal, gastrointestinal, hepatic, metabolic, endocrine, neurological or psychiatric abnormalities, and the subject is in general good health
* Subject is a nonsmoker, or has stopped smoking for at least 3 months prior to the Screening Visit
* Subject has clinical laboratory test results within the reference ranges of the laboratory. Subjects with isolated laboratory test results that are outside the reference ranges will be allowed to enroll at the discretion of the Investigator, so long as these results are deemed by the Investigator to be clinically nonsignificant
* Subject has Blood Pressure (BP) and pulse rate within normal range in supine position after 5 minutes rest (SBP: 90 to 140 mmHg, DBP: 50 to 90 mmHg, pulse rate: 45 to 100 bpm). Subjects with vital sign results that are outside the specified ranges and that are deemed clinically nonsignificant will be allowed to enroll at the discretion of the Investigator
* Subject has regular intestinal transit, in the opinion of the Investigator, determined on the basis of absence of any history or current symptoms of recurrent constipation, diarrhea, or any other gastrointestinal diseases. The mean stool frequency should be at least once every 2 days
* Subject confirms that, during the study period and for a period of 3 months after the final dose, when having sexual intercourse with a woman of childbearing potential, he will use a barrier contraceptive (eg, condom) AND that the respective partner will use an additional contraceptive method. Subject should also agree not to donate semen during this period of time

Exclusion Criteria:

* Subject has previously participated in this study or another tozadenant study
* Subject is currently participating in or has participated in another study of an investigational medicinal product or medical device in the last 3 months or 5 half-lives (whichever is longer)
* Subject has a history of exposure to ionizing radiations (except radiography) or has participated in another Absorption, Distribution, Metabolism, and Excretion (ADME) study with a radiation burden >0.1 mSv in the period of 1 year before Screening
* Subject has a history of, or present, medical or psychiatric condition that, in the opinion of the Investigator, could jeopardize or would compromise the subject's ability to participate in this study
* The subject has a known hypersensitivity to any components of the tozadenant formulation or to similar drugs (A2a antagonists), or has a history of drug or other relevant allergy that, in the opinion of the Investigator or UCB Study Physician, contraindicates their participation
* Subject has a known clinically relevant allergy or known severe adverse reaction to any drug, or known or suspected clinically relevant drug hypersensitivity that, in the opinion of the Investigator, could jeopardize or would compromise the subject's ability to participate in this study
* Subject has a history or presence of drug or alcohol dependency or tests positive for drugs or alcohol (urine tests) at Screening or Day -1
* Subject consumes more than 28 units of alcohol per week (330 mL of 5% alcohol by volume beer=2 units; 125 mL of 12% wine=1.5 units; 50 mL of 40% spirits=2 units).
* Subject consumes more than 600 mg of caffeine/ day (1 cup of coffee contains approximately 100 mg of caffeine, 1 cup of tea contains approximately 30 mg of caffeine, and 1 glass of cola contains approximately 20 mg of caffeine)
* Subject has a diet that deviates notably from the "normal" amounts of protein, carbohydrate, and fat, as judged by the Investigator (eg, vegans)
* Subject has received any prescription or nonprescription medicines, including enzyme inhibitors or inducers, over-the-counter remedies, vitamins outside the recommended daily dose limits, herbal, and dietary supplements (including St. John's Wort) within 14 days or 5 half-lives (whichever is longer) prior to administration of study medication. Occasional paracetamol use is allowed within the 14 days before the study drug administration, with a maximal dose of 2 g/day and a maximal cumulative dose of 10 g per 14 days, and during the study for the treatment of mild symptoms (eg, headache or pain relief)
* Subject has consumed any grapefruit, grapefruit juice, grapefruit containing products, or star fruit within 14 days prior to the planned administration of the study drug
* Subject tests positive for human immunodeficiency virus (HIV) -1/2 antibody (HIV-1/2 Ab), hepatitis B surface antigen (HBsAg), or hepatitis C antibody (HCV-Ab).
* Subject has a history or present condition of hepatic disorders, including but not limited to elevation of liver enzymes (alanine aminotransferase [ALT], aspartate aminotransferase [AST], alkaline phosphatase, and gamma-glutamyltransferase [GGT]) at the upper limit of laboratory reference ranges
* Subject has a history of thyroid abnormalities
* Subject has had significant blood loss or has donated or received 50 mL or more of blood within 60 days prior to drug administration, or has donated plasma or platelets within 14 days prior to first drug administration for this study
* Subject shows any sign of orthostatic hypotension at Screening, defined as:

  * A ≥20 mmHg decrease in SBP, and/or ≥10 mmHg decrease in DBP if the resultant SBP falls below 90mmHg and/or DBP falls below 60 mmHg. Blood pressure and pulse rate will be recorded after 5 minutes of rest in the supine position and after 2 minutes of rest in the standing position
  * A ≥40 mmHg decrease in SBP, and/or ≥20 mmHg decrease in DBP, regardless of resultant SBP and/or DBP. Blood pressure and pulse rate will be recorded after 5 minutes of rest in the supine position and after 2 minutes of rest in the standing position
* Subject has an abnormality in the 12-lead ECG at Screening that results, in the opinion of the Investigator, in an increase in the risks associated with participating in the study. In addition, any subject with any of the following findings will be excluded:

  * QT interval corrected for heart rate using Fridericia's formula (QTcF) >450 ms in ECG
  * Bundle branch blocks and other conduction abnormalities other than mild first degree atrioventricular block (defined as PR interval ≥220 ms)
  * Irregular rhythms other than sinus arrhythmia or occasional, rare supraventricular or ventricular ectopic beats
  * In the judgment of the Investigator, T-wave configurations are not of sufficient quality for assessing QT interval duration
* Subject has a history of unexplained syncope, or a family history of unexplained sudden death or sudden death due to long QT syndrome
* Subject has a history or present condition of respiratory or cardiovascular disorders (eg, cardiac insufficiency, coronary heart disease, hypertension, arrhythmia, tachyarrhythmia, or myocardial infarction)
* Subject has a history or present condition of malignancy, gastrointestinal bleeding, or anal fissures
* Subject is unable to understand the constraints of full urine and stool collection

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2013-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Composite of total radioactivity concentration in whole blood, plasma, urine, feces and expired air, and cumulative percentage of radioactive dose in urine and feces, and total mass balance during the study (approximately 14 days) | Samples collected during Screening Visit - Day 14 (maximum of 14 days)
  Time evolution of radioactivity in plasma, blood, urine, feces and expired air from pre-dose to day 14. Cumulative time evolution of percentage of radioactivity in urine, feces, expired air and total. Total mass balance in percentage of dose.
  This outcome measure is a composite outcome. This means that multiple measurements will be reflected as one value for each study arm.
Composite pharmacokinetic parameters of the total radioactivity during the study (approximately 14 days) | Samples collected during Screening Visit - Day 14 (maximum of 14 days)
  Pharmacokinetics parameters computed on radioactivity concentrations:
  Plasma and blood: Cmax, tmax, AUC(0-t), apparent t1/2, AUC, elimination constant (λz)
  Cumulative amount excreted in urine, feces, and expired air
  This outcome measure is a composite outcome. This means that multiple measurements will be reflected as one value for each study arm.

SECONDARY OUTCOMES:
Composite pharmacokinetic parameters of tozadenant during the study (approximately 14 days) | Samples collected during Screening Visit - Day 14 (maximum of 14 days)
  The pharmacokinetics of tozadenant in plasma and urine are evaluated using the classical set of PK parameters: Cmax, tmax, AUC(0-t), AUC, λz, t1/2, Vz/F, CL/F, Ae, fe, CLR.
  This outcome measure is a composite outcome. This means that multiple measurements will be reflected as one value for each study arm.
Identification and quantification of metabolites of tozadenant in plasma and excreta during the study (approximately 14 days) | Samples collected during Screening Visit - Day 14 (maximum of 14 days)
  For structural identification, metabolites of tozadenant in the collected HPLC fractions, using quadrupole time-of-flight mass spectrometry will be identified from plasma and excreta samples. Quantification of metabolites.

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaceutical Research Associates Group B.V., Zuidlaren, Netherlands